CLINICAL TRIAL: NCT07122362
Title: Investigation of the Effect of Elastic Lower Extremity Orthosis on Gait and Balance Parameters in Children With Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Effect of Elastic Lower Extremity Orthosis on Gait and Balance in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ERKAN, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024 - 587
Record Dates: First submitted 2025-07-30; First posted 2025-08-14 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Spastic Cerebral Palsy
Keywords: cerebral palsy; in-toeing gait; balance; orthoses; neoprene
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Neurodevelopmental Therapy (Active Comparator): Participants receive conventional neurodevelopmental therapy only.
  Interventions: Behavioral: Neurodevelopmental Therapy
- Intervention Group: Therapy + Elastic Orthosis (Experimental): Participants receive conventional neurodevelopmental therapy plus elastic lower extremity orthosis.
  Interventions: Device: Elastic Lower Extremity Orthosis; Behavioral: Neurodevelopmental Therapy

INTERVENTIONS:
Device: Elastic Lower Extremity Orthosis — Participants in the intervention group receive conventional neurodevelopmental therapy combined with an elastic lower extremity orthosis designed to correct internal rotation deformities and improve gait and balance in children with spastic cerebral palsy. The orthosis applies elastic tension around the femoral region and tibia to target rotational problems.
  Arms: Intervention Group: Therapy + Elastic Orthosis
Behavioral: Neurodevelopmental Therapy — Participants receive conventional neurodevelopmental therapy only.

SUMMARY:
This randomized controlled trial aims to evaluate the effect of an elastic lower extremity orthosis on gait and balance in children with spastic cerebral palsy who present with an in-toeing gait pattern. The study compares conventional neurodevelopmental therapy alone to therapy combined with the orthosis.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of permanent disorders affecting movement and posture and is one of the most common causes of motor disability in children. One of the most frequent rotational gait abnormalities in children with spastic CP is in-toeing, which may result from increased femoral anteversion, internal tibial torsion, or foot deformities such as metatarsus varus or metatarsus adductus.

Elastic orthoses wrapped around the femoral region can generate active rotational forces and help modify the foot progression angle during gait. In early childhood, elastic external rotation straps starting from the foot can also be used for tibial rotation problems.

This randomized controlled trial will compare the effects of conventional neurodevelopmental therapy alone with therapy combined with the use of an elastic lower extremity orthosis.

Primary outcome measure: Gait parameters

Secondary outcome measure: Balance parameters

The study hypothesizes that the group receiving the orthosis in addition to conventional therapy will demonstrate superior outcomes in terms of gait and balance compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation
* Diagnosis of spastic cerebral palsy
* Gross Motor Function Classification System (GMFCS) level 1, 2, or 3
* Age between 18 and 84 months
* Presence of in-toeing gait pattern

Exclusion Criteria:

* GMFCS level 4 or 5
* Botulinum toxin injection or surgical intervention targeting the lower extremities or pelvis within the last 6 months

Ages: 18 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Gait parameters assessed by Edinburgh Visual Gait Analysis | Baseline and 8 weeks after intervention
  The Edinburgh Visual Gait Analysis Scale will be used to assess changes in gait patterns before and after the intervention. This scale consists of 17 items. Each item is scored between 0 and 2. A total score closer to zero indicates improved gait. The Edinburgh Visual Gait Analysis Scale was developed to quantitatively analyze gait parameters at different stages in recorded videos. During the assessment, children will be videotaped walking on a flat surface with their lower extremities bare. These recordings will assess each lower extremity during the stance and swing phases of gait.

SECONDARY OUTCOMES:
Balance parameters assessed by Pediatric Balance Scale | Baseline and 8 weeks after intervention
  The Pediatric Balance Scale will be used to assess balance performance and changes in balance ability at baseline and 8 weeks after the intervention. The 14-item Pediatric Balance Scale is a functional balance measurement tool adapted for the pediatric population and allows for the assessment of balance in various positions and during movement; each item is scored from 0 to 4, with the highest possible score being 56. A higher score indicates better balance.

CONTACTS AND LOCATIONS:
Overall Officials: BÜLENT ELBASAN, Prof., Study Chair — Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Gazi University, Ankara, Türkiye
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Gazi University, Ankara, Turkey, Ankara, Ankara
  - Niğde Ömer Halisdemir University Bor Physical Therapy and Rehabilitation Training and Research Hospital, Niğde, Niğde Province

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request from qualified researchers with ethics approval, starting 6 months after study completion. Data sharing will be conducted under a data sharing agreement to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data and supporting documents will be available starting 6 months after study completion and will remain available for at least 5 years.
Access Criteria: Qualified researchers with appropriate ethics committee approval may request access to the de-identified IPD and supporting documents. Data will be shared following a data sharing agreement that ensures confidentiality and appropriate use. Access requests can be made by contacting the corresponding

DOCUMENTS (2):
  • Study Protocol (2025-04-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT07122362/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT07122362/SAP_001.pdf